CLINICAL TRIAL: NCT02165228
Title: A Stress Reduction Strategy for Decreasing CVD Risk Through C-reactive Protein Reduction
Brief Title: Strategies for Inflammation and Cardiovascular Disease (CVD) Prevention
Acronym: SICVDP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Mary Miles, Professor, Montana State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10GRNT260013
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Atherosclerosis; Diabetes
MeSH Terms: conditions — Atherosclerosis; Diabetes Mellitus | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mindfulness-based stress reduction (Experimental): Stress reduction class and behavioral intervention
  Interventions: Behavioral: Mindfulness-based stress reduction
- Nutrition Enhancement (Active Comparator): Nutrition education class and behavioral intervention
  Interventions: Behavioral: Nutrition Enhancement
- Control (No Intervention): No class or behavioral intervention

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction — Stress reduction class and behavioral intervention
  Arms: Mindfulness-based stress reduction
Behavioral: Nutrition Enhancement — Nutrition education class and behavioral intervention
  Arms: Nutrition Enhancement

SUMMARY:
The long-term goal of the proposed research is to identify and develop effective interventions to decrease persistent, low-level inflammation and risk of CVD. Stress is a substantial contributor to inflammation, and interactions among stress, inflammation, body mass index, and health behaviors have been measured. Mindfulness-based stress reduction (MBSR) is effective for stress reduction, has been shown to be effective for inflammation reduction in individuals with disease, and is a sustainable practice for individuals across the health spectrum. Diet strategies are an effective means of reducing inflammation for some individuals, but may not be successful for many people, as evidenced by the steady rise in obesity rates. The specific aims of this study are to 1) test the effectiveness of MBSR compared to an established intervention of a nutrition enhancement (NE) intervention for the reduction of inflammation, and 2) test the effectiveness of MBSR compared to a non-intervention control conditions (CON) for the reduction of inflammation. Men and women 25-45 years of age will be randomly assigned to participate in MBSR (n=60) or DIET (n=60) or CON (n=60) interventions for 16 weeks. Serum CRP concentrations, additional inflammatory cytokines (tumor necrosis factor-a, interleukin-6), cortisol diurnal profiles, anthropometrics, dietary intake, and all components of the metabolic syndrome will be measured pre- and post-intervention to elucidate underlying mechanisms and to determine whether health benefits beyond inflammation reduction occur.

ELIGIBILITY:
Inclusion Criteria:

* Elevated waist circumference or BMI

Exclusion Criteria:

* Participation in calorie restricted diet in previous 30 d
* Participation in stress reduction program in previous 30 d
* Take blood pressure, lipid lowering or anti-inflammatory medications
* Hypertension
* Diabetes
* Heart disease

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2010-01; Primary Completion 2012-03 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Inflammation Biomarkers | 16 weeks
  C-reactive protein (CRP), tumor necrosis factor-alpha, interleukin-6
Metabolic Syndrome Extent | 16 weeks
  Blood pressure, waist circumference, fasting glucose, fasting HDL, fasting triglycerides, number of components

SECONDARY OUTCOMES:
BMI | 16 weeks
  BMI = weight/height squared
Waist to hip ratio | 16 weeks
  Circumference of the waist/circumference of the hips
Cholesterol | 16 weeks
  Fasting total cholesterol concentration
Insulin Resistance | 16 weeks
  Fasting insulin concentration and homeostatic model assessment of insulin resistance (HOMA-IR)
Stress hormone levels | 16 weeks
  Salivary cortisol concentration at 7 a.m., 12 and 4 p.m.
Perceived Stress | 16 weeks
  Score from the perceived stress scale.
Depression | 16 weeks
  Depression Score
Mindfulness | 16 weeks
  Perception of mindfulness from subscale within the self-compassion scale questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mary P Miles, PhD, Principal Investigator — Montana State University
Locations (1):
- Montana State University, Bozeman, Montana, United States